CLINICAL TRIAL: NCT01726153
Title: A Pilot Randomized Control Trial (RCT) of an Individualized Condom-HIM Web-based Intervention for Condom USe Among HIV+ Gay Males
Brief Title: A Pilot Trial of an Individualized Web-Based Condom Use Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R0018767
Record Dates: First submitted 2012-11-06; First posted 2012-11-14 (Estimated); Last update posted 2020-07-24 (Actual); Status verified 2012-11

CONDITIONS: HIV
Keywords: Condom Use; HIV+ gay males; Intervention; Tailored; On-line; Internet; Web-based

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Web sites (No Intervention): Individuals assigned to this arm are given a list of websites where they can view additional information relating to condom use.
- Condom-HIM (Experimental): Individuals assigned to this arm must follow an on-line one session tailored intervention.
  Interventions: Behavioral: Condom-HIM

INTERVENTIONS:
Behavioral: Condom-HIM — The tailored on-line Condom-HIM intervention is composed of a single session involving activities to increase individuals self-efficacy and intention to use condoms.
  Arms: Condom-HIM

SUMMARY:
The purpose of this study is to evaluate the efficacy of an online intervention in increasing condom use among HIV+ gay males.

ELIGIBILITY:
Inclusion Criteria:

1. are HIV-seropositive,
2. Men who are having sex with men,
3. engaging in unprotected anal intercourse with a partner who is serostatus negative or unknown
4. age 18 years and older,
5. ability to read English
6. have access to a computer and internet.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-11; Primary Completion 2013-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in participants self-efficacy in condom use at 2-weeks post-intervention | baseline and 2-weeks post intervention
  The Self-Efficacy for condom use measure contains a set of items to rate participant's belief that they will be able to use condoms every time they have anal sex in a variety of situations. A four-point response scale, ranging from 'strongly agree' (0) to 'strongly disagree' (4) is used. The psychometric properties of the measure have been examined and have been shown to have good internal consistency with Cronbach's alpha coefficient of 0.96.

SECONDARY OUTCOMES:
Change from Baseline in participants intention to use condoms at 2-weeks post-intervention | Baseline and 2-weeks post intervention
  The intention to use condoms measure asks participants their intention to consistently use condoms. The psychometric properties of the measure have been examined and have shown to have good internal consistency with Cronbach's alpha coefficient of 0.89.

OTHER OUTCOMES:
Change from Baseline in participants condom use at 2-weeks post-intervention Condom Use | baseline and 2-weeks post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Joyal Miranda, PhD, Principal Investigator — Ryerson University and Centre hospitalier de l'Universite de Montreal (CHUM)
Locations (1):
- Ryerson University, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Miranda J, Cote J, Godin G, Blais M, Otis J, Gueheneuc YG, Fadel G, Barton L, Fowler S. An Internet-Based Intervention (Condom-Him) to Increase Condom Use Among HIV-Positive Men Who Have Sex With Men: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2013 Oct 16;2(2):e39. doi: 10.2196/resprot.2723. PMID 24132072